CLINICAL TRIAL: NCT00458380
Title: Clinical Use of the Perifollicular Vascularity Assessment in in-Vitro Fertilization Cycles: a Pilot Study
Brief Title: Perifollicular Vascularity Assessment in in-Vitro Fertilization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 09/2004
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Last update posted 2007-04-10 (Estimated); Status verified 2007-04

CONDITIONS: Infertility
Keywords: Doppler ultrasonography; Embryos; Infertility; IVF; Oocytes; Tubal factor; unexplained infertility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Controlled ovarian stimulation, perifollicular vascularity assessment, IVF, embryo transfer.

SUMMARY:
On February 2004, a law (n. 40/2004) regulating assisted reproduction techniques (ARTs) was approved in Italy. This law aimed to regulate the treatment of infertility in Italy, contains several restrictions, such as the prohibition to fertilize more than three oocytes and the obligation to transfer simultaneously all embryos obtained. Several evidences showed that the outcome of the in-vitro fertilization (IVF) techniques is strongly correlated with quality of transferred embryos (choosing the right embryos). Furthermore, this prerequisite is actually illegal in Italy, and an optimal oocyte selection can be considered as the only one crucial factor in the determining the outcome of the IVF cycle (choosing the right oocytes). Experimental data have demonstrated that perifollicular blood flow assessment is a good marker of oocyte competence, embryo viability, implantation potential, and subsequent pregnancy rate.

The purpose of this study will be to evaluate in a clinical setting whether the assessment of the perifollicular vascularity is a feasible and useful procedure for the selection of oocytes with the best developmental potential in IVF programs when only a limited number of oocytes can be fertilized.

DETAILED DESCRIPTION:
One hundred fourteen women with tubal factor or unexplained infertility undergoing IVF programs in our department will be enrolled in a wild protocol. Successively, the enrolled patients will be divided into two different sub-protocols evaluating the role of the perifollicular vascularity in good- and poor-prognosis patients. The diagnosis will be established by hysterosalpingography and/or laparoscopic dye test and with partner's semen analysis.

All patients will be randomly allocated in two independent groups (experimental and control groups) using a computer-software, and the random allocation sequence will be concealed in closed and dark envelope until the interventions will be assigned.

In the experimental group alone, a power Doppler assessment of perifollicular vascularity will be performed the day of oocyte retrieval (36 h after hCG injection). The vascularity of each ovulatory follicle will be successively studied using an advanced image analysis software and its extension will be graded using a well validated grading system. The periovulatory follicles will be categorized in high-grade (grades 3-4) and low-grade (grades 1-2).

After patient' sedation with IV propofol, oocytes will be retrieved using a 17 G double-lumen aspiration needle with a low pressure and individually cultured marking the test-tube and, successively, the culture plate with a code corresponding to perifollicular vascularity degree. The retrieved oocytes will be washed and the mature oocytes, determined by the presence of a first polar body (metaphase II; MII oocytes), will be classified by an experienced biologist initially blinded to previous perifollicular vascularization. In particular, MII oocytes will be graded into three groups according to the number of anomalies: grade I, oocytes without any anomaly; grade II, oocytes with one anomaly; and grade III, oocytes with at least two anomalies.

The three oocytes with the highest grade will be considered "the best" oocytes to fertilize in the control group, whereas in the experimental group they will be selected integrating morphological and ultrasonographic criteria. In particular, the embryologist will use the ultrasonographic criteria to choice within oocytes with similar morphologic degree.

In both groups, three MII oocytes will be inseminated at 4 h after recovery with 10000-20000 motile sperm and placed in the CO2 incubator at a temperature of 37°C in 5% CO2 in air, and the fertilization will be evaluated 18 h later and confirmed by the presence of two pronuclei and two polar bodies. The fertilized oocytes will be classified with a well standardized scoring system for zygotes and cultured for a total of 48 h from oocytes IVF. Before transfer, the cleavage embryos will be again graded according to the embryo morphology and the relative proportion of anucleate fragments present in the zona pellucida.

All embryos, with exclusion of those arrested (not cleaved after 24 h from IVF), will be replaced in each patient without ultrasonographic guidance using ultrasoft Frydman catheter. The luteal phase will be supported by 100 mg natural progesterone daily administrated. A serum β-hCG assessment will be performed on 15th day after embryos transfer.

For each cycle, the serum estradiol levels and the number of dominant follicles on the day of hCG administration, the duration of ovarian stimulation, and the units of r-FSH administered will be recorded. The concordance between the ultrasonographic grading score and the oocyte degree will be also evaluated in each case.

Cancelled cycles (cases of absence of follicular response after 35 days of treatment or a serum E2 value >2500 pg/ml), fertilization (percentage of fertilized oocytes / total oocytes), implantation (percentage of intra-uterine gestational sacs / total transferred embryos), clinical (percentage of rising β-hCG with sonographic evidence of intrauterine gestational sac and fetal cardiac activity at 7 weeks of pregnancy / total non-cancelled cycles) and ongoing (percentage of vital pregnancies confirmed by ultrasonography at 12 weeks of gestational age / total non-cancelled cycles) pregnancies rates will be evaluated in each patients. The number of multiple pregnancies and ovarian hyperstimulation syndromes (OHSS) will be also recorded in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with tubal factor or unexplained infertility undergoing IVF programs.

Exclusion Criteria:

* Body mass index (BMI, Kg/m2) <18 and >30
* Peritoneal factor infertility
* Polycystic ovaries (PCO)
* Other organic pelvic diseases
* Abnormal partner's semen
* Neoplastic, metabolic, endocrinological, hepatic, and cardiovascular disorders or other concurrent medical illness
* Abuse of alcohol
* Current or previous use of hormonal drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116
Dates: Start 2004-09; Study Completion 2005-02

PRIMARY OUTCOMES:
Ongoing pregnancy rate

SECONDARY OUTCOMES:
Implantation rate

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy

REFERENCES:
- [Result] Palomba S, Russo T, Falbo A, Orio F Jr, Manguso F, Nelaj E, Tolino A, Colao A, Dale B, Zullo F. Clinical use of the perifollicular vascularity assessment in IVF cycles: a pilot study. Hum Reprod. 2006 Apr;21(4):1055-61. doi: 10.1093/humrep/dei441. Epub 2005 Dec 22. PMID 16373407